CLINICAL TRIAL: NCT06898359
Title: Role of Gut Microbiota in Neoadjuvant Radioimmunotherapy for MSS, Locally Advanced Rectal Cancer: A Single-Center, Observational Study
Brief Title: Role of Gut Microbiota in Neoadjuvant Radioimmunotherapy for MSS, Locally Advanced Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: GIHSYSU-SAH-01
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; PD-1; micobe
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radioimmunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We have collected the feces, serum and colonoscopy biopsy specimens of the patients before treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radioimmunotherapy — SCRT (a total of 25 Gy in 5 days) followed by sintilimab (3mg/kg intravenous drip on day 1; every 3-week cycle for two cycles)

SUMMARY:
This research investigates the role of the gut microbe in patients receiving radioimmunotherapy with locally advanced microsatellite-stable (MSS) rectal cancer. Given the limitations of current treatment strategies in achieving optimal clinical outcomes, this prospective, single-center, phase II clinical trial aims to improve pathological complete response (pCR) rates. The primary endpoint is pCR, with secondary endpoints including disease-free survival (DFS) and the incidence of treatment-related adverse events. This study seeks to provide insights into a novel treatment paradigm for MSS locally advanced rectal cancer, potentially offering improved therapeutic options for this patient population.

DETAILED DESCRIPTION:
Locally advanced rectal cancer (LARC) presents a complex treatment challenge, often requiring a multimodal approach to achieve optimal cure rates and improve survival. Currently, the combination of short-course radiotherapy (SCRT) and neoadjuvant chemotherapy has become a critical treatment strategy for LARC patients. Compared to conventional long-course radiotherapy (LCRT), SCRT is associated with a shorter treatment duration, typically lasting only five days, which facilitates rapid tumor shrinkage and minimizes surgical delays. This expedited treatment approach not only reduces the risk of postponing surgery but also improves the management of patients by minimizing fatigue and treatment-related side effects associated with longer regimens.

Despite the promising outcomes associated with SCRT and neoadjuvant chemotherapy, a significant proportion of patients still do not achieve satisfactory clinical responses to standard treatment regimens.

In recent years, the emergence of immune checkpoint inhibitors has revolutionized cancer treatment. In particular, PD-1 inhibitors such as Sintilimab have demonstrated significant antitumor activity across various solid tumors, notably in microsatellite instability-high (MSI-H) cancers. However, the potential benefits of these agents in microsatellite-stable (MSS) rectal cancer remain insufficiently explored.

This study aims to investigate the effects of radioimmunotherapy in a single-center cohort for MSS locally advanced rectal cancer. We hope to provide a novel therapeutic option that enhances clinical efficacy for patients with LARC by evaluating the differences in the gut microbiota in those patients with pCR vs no-pCR response.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

With my consent and signed informed consent, willing and able to comply with the planned visit, research treatment, laboratory tests, and other test procedures; Age 18-75; Patients with a pathologically or cytologically confirmed adenocarcinoma of the rectum, all other histological types excluded; The distance between the lower margin of the rectal tumor lesion and the anal margin <12cm; The physical status score (ECOG) of the Eastern United States Cancer Cooperative Group was 0-1 (see Appendix 1); T3-4/N+ was evaluated by pelvic enhanced MRI; Had not received systemic anti-tumor therapy for colon cancer, including cytotoxic drugs, immune checkpoint inhibitor therapy, molecular targeted therapy, endocrine therapy, etc.; Appropriate organ function based on the following laboratory test values obtained during the screening period: White blood cell count ≥3×109/L, neutrophil count ≥1.5×109 /L, platelet count ≥75×109 /L, serum total bilirubin ≤ 1.5× upper limit of normal (UNL), AST (SGOT) or ALT (SGPT) ≤ 2.5×UNL, serum creatinine ≤ 1.5×UNL; Female subjects of reproductive age must undergo a negative serum pregnancy test within 3 days prior to the start of the study drug and be willing to use a medically approved highly effective contraceptive method (such as an IUD, contraceptive pill, or condom) during the study period and within 3 months after the last study drug administration; Male subjects whose partners are women of reproductive age should be surgically sterilized or agree to use effective contraception during the study period and for 3 months after the last study dosing; Willing and able to comply with research procedures and visit plans.

Exclusion Criteria:

Whole-body CT, MR, or PET-CT (including at least the chest, whole abdomen, and pelvis) confirms distant metastases (M1); Patients with complete intestinal obstruction, active bleeding or perforation requiring emergency surgery; The presence of other active malignancies in the past or at the same time (except malignancies that have received curative treatment and have been free of disease for more than 5 years or cancers in situ that can be cured by adequate treatment); Thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, and deep vein thrombosis, occurred in the 12 months before study entry; Myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac dysfunction, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure in the 12 months prior to enrollment; Systemic antibiotic use ≥ 7 days within 4 weeks prior to enrollment, or unexplained fever &gt during screening/prior to first dosing; 38.5°C (as determined by the investigators, fever due to tumor could be included); Had received major operations such as laparotomy, thoracotomy, laparoscopic resection of organs or severe trauma within 2 months before enrollment (the surgical incision should be completely healed before enrollment in this clinical trial); Known presence of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) related disease; The presence of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases (such as diabetes, hypertension, pulmonary fibrosis and acute pneumonia); Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; Hepatitis C, defined as HCV-RNA above the lower detection limit of analytical methods) or co-infection with hepatitis B and hepatitis C; A known or suspected history of allergy to any of the relevant drugs used in the study; Pregnant or lactating women; Women of reproductive age who do not use or refuse to use effective non-hormonal contraception (after the last menstrual period < 2 years) or men who are likely to have children; The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participating in the study or interfere with the study results, as well as patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with MSS Locally Advanced Rectal Cancer following Locally Advanced Rectal Cancer
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Pathological complete response | 1 month after the surgery]
  Pathological complete response will be evaluated with the American Joint Committee on Cancer (AJCC) Cancer Staging

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital of Sun yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No